CLINICAL TRIAL: NCT05887804
Title: Comparison of Keloid Volume and Symptoms Reduction Between Intralesional Umbilical-Cord Mesenchymal Stem Cells, Its Conditioned Medium, and Triamcinolone Acetonide Injection as Keloid Therapy: A Randomised Controlled Trial
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Rumah Sakit Pusat Angkatan Darat Gatot Soebroto (Other)
Collaborators: Indonesia University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KET-1206
Record Dates: First submitted 2023-05-24; First posted 2023-06-05 (Actual); Last update posted 2023-06-07 (Actual); Status verified 2023-06

CONDITIONS: Keloid; Stem Cell
Keywords: Keloid therapy; mesenchymal stem cells; keloid volume; POSAS
MeSH Terms: conditions — Keloid | interventions — Triamcinolone Acetonide

STUDY DESIGN:
Intervention Model Description: Patients were screened initially by measuring the length and thickness of the keloids using a ruler. Patients who met the study inclusion criteria were randomly divided into 3 groups. Each patient in the groups was given the same injection volume (1 mL) in every cm3 keloid volume using a 1 mL syringe and 27G needle. The injections were ultrasound-guided into the center of the lesion with a 30-45-degree angle using an in-plane technique, therefore the same pressure. Group 1 was given UC-MSC 2 million cells/mL/cm3, group 2 was given UC-CM 1 mL/cm3, and group 3 was given TA 40 mg/mL/cm3.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The laboratory staff prepared the substances in identical syringes without informing the researchers according to randomization. Data processing was carried out by statisticians and clinicians other than researchers.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- umbilical cord-derived mesenchymal stem cells (UC-MSC) (Experimental): UC-MSC was collected in 50 mL of transport medium, which contained alpha minimal essential medium (αMEM [GIBCO 12000-0221]), penicillin/streptomycin (final concentration 300u/mL [GIBCO 15140-122]) and amphotericin B (final concentration 7500ng /mL [JR Scientific 50701]), and processed in less than 8 hours after collection.
  Group 1 was given UC-MSC 2 million cells/mL/cm3
  Interventions: Biological: umbilical cord-derived mesenchymal stem cells (UC-MSC)
- umbilical cord-derived mesenchymal stem cells conditioned medium (UC-CM) (Experimental): group 2 was given UC-CM 1 mL/cm3
  Interventions: Biological: umbilical cord-derived mesenchymal stem cells conditioned medium (UC-CM)
- triamcinolone acetonide (Active Comparator): group 3 was given TA 40 mg/mL/cm3
  Interventions: Drug: Triamcinolone Acetonide (TA)

INTERVENTIONS:
Biological: umbilical cord-derived mesenchymal stem cells (UC-MSC) — Group 1 was injected UC-MSC 2 million cells/mL/cm3, given the same injection volume (1 mL) in every cm3 keloid volume using a 1 mL syringe and 27G needle. The injections were ultrasound-guided into the center of the lesion with a 30-45-degree angle using an in-plane technique, therefore the same pressure.
  Arms: umbilical cord-derived mesenchymal stem cells (UC-MSC)
Biological: umbilical cord-derived mesenchymal stem cells conditioned medium (UC-CM) — Group 2 was injected UC-CM 1 mL/cm3, given the same injection volume (1 mL) in every cm3 keloid volume using a 1 mL syringe and 27G needle. The injections were ultrasound-guided into the center of the lesion with a 30-45-degree angle using an in-plane technique, therefore the same pressure.
  Arms: umbilical cord-derived mesenchymal stem cells conditioned medium (UC-CM)
Drug: Triamcinolone Acetonide (TA) — Group 3 was injected TA 40 mg/mL/cm3, given the same injection volume (1 mL) in every cm3 keloid volume using a 1 mL syringe and 27G needle. The injections were ultrasound-guided into the center of the lesion with a 30-45-degree angle using an in-plane technique, therefore the same pressure.
  Arms: triamcinolone acetonide

SUMMARY:
This study is a double-blind randomized controlled trial (RCT) examining the effect of intralesional injection of umbilical cord-derived mesenchymal stem cells (UC-MSC), umbilical cord-derived conditioned medium (UC-CM), or triamcinolone acetonide (TA) on keloids carried out using CONSORT statement. Research is directed at studying keloid volume reduction and changes in POSAS score.

DETAILED DESCRIPTION:
Patients were screened initially by measuring the length and thickness of the keloids using a ruler. Patients who met the study inclusion criteria were randomly divided into three groups. Each patient in the groups was given the same injection volume (1 mL) in every cm3 keloid volume using a 1 mL syringe and 27G needle. The injections were ultrasound-guided into the center of the lesion with a 30-45-degree angle using an in-plane technique, therefore the same pressure. Group 1 was given umbilical cord-derived mesenchymal stem cells (UC-MSC) 2 million cells/mL/cm3, group 2 was given umbilical cord-derived conditioned medium(UC-CM) 1 mL/cm3, and group 3 was given triamcinolone acetonide (TA) 40 mg/mL/cm3. All patients received a single dose and 1 booster dose. The percentage of keloid volume regression in each treatment group was calculated by calculating the difference in volume before and after therapy with a 3-dimensional CT-scan, then expressed as a percentage. The CT-scan volume was obtained with the SmartVitrea application (Figure 2), then a POSAS examination will be carried out for subjective and objective assessment.

ELIGIBILITY:
Inclusion Criteria:

* The patient has keloids with a length of 2-10 cm and a thickness of 3-5 mm located on the chest, back, abdomen and extremities
* Patients aged 18 - 55 years
* Post-surgery patients more than 3 months that cause keloids
* The patient is willing to fill in the informed consent form

Exclusion Criteria:

* Patients with hypertrophic scars
* History of kidney failure
* Hypertension
* Pregnant and breastfeeding
* History of blood disorders
* History of tumor or malignancy
* Get other keloid therapy outside of the research procedure

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-06-09 (Actual); Study Completion 2022-06-09 (Actual)

PRIMARY OUTCOMES:
Keloid volume reduction | 15 weeks
  Volume was measured by CT-scan 2 weeks and 17 weeks after the first visit
The Patient and Observer Scar Assessment Scale (POSAS) score reduction | 17 weeks
  Symptoms were measured using The Patient and Observer Scar Assessment Scale (POSAS) on the first visit, five weeks, 13 weeks, and 17 weeks after the first visit. Each item of the POSAS is rated on a 10-point score. The lowest score is '1', corresponding to the normal skin situation (i.e., normal pigmentation, no itching). Score 10 equals the most significant difference from normal skin (i.e., the worst imaginable scar or sensation). The symptoms are considered improved if the score gets lower. The total score of both scales can be calculated by summing up the scores of each of the six items. The total score can range from 6 to 60.

CONTACTS AND LOCATIONS:
Locations (1):
- RSPAD Gatot Soebroto, Jakarta Pusat, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: No